CLINICAL TRIAL: NCT02653755
Title: The PRECISION Trial (Profiling Early Breast Cancer for Radiotherapy Omission): A Phase II Study of Breast-Conserving Surgery Without Adjuvant Radiotherapy for Favorable-Risk Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: NanoString Technologies, Inc. (Industry)
Responsible Party: Principal Investigator, Julia S. Wong, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-255
Record Dates: First submitted 2016-01-10; First posted 2016-01-12 (Estimated); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer Radiation
Keywords: Breast Cancer Radiation; Radiotherapy for Favorable-Risk Breast cancer; Radiotherapy Omission

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Ineligible for omission of RT (Active Comparator): Prosigna confirms intermediate- or high-risk score. Participants with intermediate- or high-risk scores will be ineligible for omission of radiotherapy (RT). Some patients with low-risk scores may elect to receive RT.
  Interventions: Device: Prosigna
- Eligible for omission of RT (Active Comparator): Prosigna confirms low risk score. Participant will be eligible for omission of therapy and chooses to do so. Patient will receive adjuvant endocrine therapy.
  Interventions: Device: Prosigna

INTERVENTIONS:
Device: Prosigna — Transcriptional profile of 50 genes used for risk stratification.
  Other Names: PAM-50

SUMMARY:
This research study is a way of gaining new knowledge about whether patients can omit radiation treatment after undergoing a lumpectomy, also known as "breast conserving surgery". In this trial, we are attempting to identify which patients may not need radiation.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational treatment to learn whether it is appropriate for treating a specific disease.

The purpose of this study is to determine whether certain patients between the ages of 50 and 75 can safely omit radiation treatment after having a lumpectomy.In this research study, the investigators are using standard laboratory tests along with the Prosigna test to see if certain patients can avoid radiation, without having a higher risk of the cancer coming back in the future.

A portion of the participant surgical specimen will be prospectively maintained for future study using institutionally-approved tissue banking procedures.

The FDA (the U.S. Food and Drug Administration) has cleared the Prosigna test for generating a risk category and numerical score to assess the risk of distant recurrence, and has cleared us to investigate the use of the Prosigna test for helping with decisions about radiation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive breast cancer
* The primary tumor must be excised via breast conserving surgery ("lumpectomy") with negative margins ("no ink on tumor") or re-excision showing no residual disease in the re-excision specimen.
* The tumor must be ≤2 cm (T1) in the largest dimension.
* Immunohistochemical studies must demonstrate the tumor to be ER+ (≥10%) or PR+, HER2- and grade 1 or 2.
* The patient must have undergone either sentinel lymph node biopsy (SLNB) or axillary lymph node dissection (ALND) demonstrating pathologic node-negativity (pN0). However, patients with immunohistochemical evidence of isolated tumor cells in a lymph node [pN0(i+)] are eligible if no deposit >0.2mm is identified.
* Age: this study is open to patients between 50 and 75 years of age (inclusive). Patients younger than 50 years of age are excluded based on prior data suggesting a different natural history for breast cancers arising in premenopausal women (with different subtype and biologic distributions that may confound the current aims). Women older than 75 years of age are excluded from this protocol due to historical difficulties achieving robust follow-up in this population, along with competing comorbidities which have been shown to interfere with subsequent breast cancer monitoring and evaluation.
* ECOG performance status ≤2 (Karnofsky ≥60%)
* Life expectancy of >5 years per the clinical impression of the treating physician(s).
* Eligible for and willing to undergo a course of adjuvant endocrine therapy.

Exclusion Criteria:

* At the time of enrollment, subjects may not have had any prior systemic therapy for breast cancer, including chemotherapy, hormonal therapy or targeted biologic therapy. Similarly, chemotherapy or biologic therapy must not be part of the subsequent treatment plan.
* Clinical, radiographic or pathologic evidence of multicentric disease.
* Evidence of T4 disease (e.g., involvement of the chest wall, skin, dermal lymphatics, or inflammatory breast cancer).
* Grade 3 histology.
* Tumors in which the invasive component is present only as micro-invasion.
* Multicentric invasive or in site carcinoma
* Bilateral breast malignancy.
* Inability or unwillingness to tolerate endocrine therapy.
* Documented mutation of TP53, BRCA1, BRCA2, or other hereditary cancer syndromes.
* Significant comorbidity associated with an estimation of <5 remaining life years.
* Another diagnosis of malignancy within the 5 years preceding enrollment (excluding non-melanoma skin cancers or in situ cervical lesions, which are permitted).
* Inability to understand or provide informed consent.
* Current addictive or psychiatric disorder which may preclude protocol adherence.
* Prior breast or chest radiotherapy for any indication.
* Pregnant or lactating.

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 671 (Actual)
Dates: Start 2016-05; Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Five-Year Risk of Local Regional Recurrence in the Ipsilateral Breast or Lymph Nodes in Women without Adjuvant Radiotherapy | 5 years
  Using information gathered from follow-up physical examinations and mammography, the 5-year risk of local regional recurrence in women who omit radiotherapy post-lumpectomy will be evaluated.

SECONDARY OUTCOMES:
Five-Year Risk of Any Recurrence: Local, Regional or Distant | 5 years
  Using information gathered from follow-up physical examinations and mammography, the 5-year risk of any recurrence in women who omit radiotherapy post-lumpectomy will be evaluated.
Overall Survival | 5 years
  Using information gathered from follow-up appointments and other record sources, 5-year survival rates will be evaluated.
Disease-Free Survival | 5 years
  Using information gathered from follow-up physical exams, mammography and other imaging as necessary, the rate of disease-free status at 5 years will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Wong, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (6):
- United States (6):
  - Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - NYU Langone Health, New York, New York
  - Memorial Sloane Kettering Cancer Center, New York, New York
  - Lifespan Cancer Institute, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ho AY, Bellon JR. Overcoming Resistance - Omission of Radiotherapy for Low-Risk Breast Cancer. N Engl J Med. 2023 Feb 16;388(7):652-653. doi: 10.1056/NEJMe2216133. No abstract available. PMID 36791166